CLINICAL TRIAL: NCT04011839
Title: Evaluation of Perineural Catheterization Practices in Postoperative Orthopedic Surgery
Acronym: Cathepos
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: Local/2018/JL-01
Record Dates: First submitted 2019-07-02; First posted 2019-07-09 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Levobupivacaïne — Use of Levobupivacaïne instead ropivacaïne

SUMMARY:
Continuous peripheral nerve blocks are considered as the gold standard for postoperative analgesia in orthopaedic surgery (shoulder, knee, foot). These techniques are also used in chronic pain.

The main disadvantage of these techniques is that they can drive a more or less deep motor block that slows down the rehabilitation process. This disadvantage could be prevented (or minimized) by adapting the protocol for administering local anesthetics or by changing molecules (levobupivacaine 0.625 mg/ml instead of ropivacaine 2 mg/ml). There is no literature comparing the effectiveness of the sensory block and its impact on the motor block according to the administration protocol and/or the type of local anesthetics.

The main judgement criterion of such a study could be a composite criterion crossing the quality of the sensory block and the depth of the motor blockades, the ideal being to have a perfect sensory block without any motor block.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* ASA score 1 to 4
* Scheduled orthopaedic surgery
* consent to participate

Exclusion Criteria:

* Pregnant, parturient, or breastfeeding woman
* Emergency situation
* Contraindications to local anaesthesia
* Patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients undergoing scheduled orthopedic surgery for which perinervous catheter analgesia is usually indicated (complex shoulder, elbow, femur, knee, foot surgery) will be included.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2022-06-29 (Actual); Study Completion 2022-06-29 (Actual)

PRIMARY OUTCOMES:
Comparison between sensory Block Quality and motor Block deep | Day1 to Day 3
  Composite score between 0 to 2 for Sensory Block and 0 to 2 for motor Block

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de NIMES, Nîmes, France

IPD SHARING:
Plan to Share IPD: Undecided